CLINICAL TRIAL: NCT02522585
Title: Predictive Value of p16 and Ki-67 Immunohistochemical Staining and NK Cells in Expectant Management of Cervical Intraepithelial Neoplasia Grade 2
Brief Title: p16 and Ki-67 Stainings and Natural Killer (NK) Cells in CIN-II Management
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Jordi Genoves, MD, PhD, Parc de Salut Mar
Other Study IDs: CIN-II p16 NK
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Cancer
Keywords: expectant management; p16; immunohistochemistry; regression; progression; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Disease Progression; Uterine Cervical Dysplasia | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Citologies and biopsies of the cervix. Blood cells.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Conservative management: Patients diagnosed of CIN-II by directed biopsy
  Interventions: Other: Conservative management

INTERVENTIONS:
Other: Conservative management — Control of CIN-II with cytology and colposcopy to try to avoid unnecessary surgery

SUMMARY:
The objective of this study is to evaluate the outcome of cervical intraepithelial neoplasia grade 2 (CIN-II) patients followed up without treatment for 24 months according to p16 and ki-67 immunohistochemical staining and to the expression of NK cell receptors.

DETAILED DESCRIPTION:
Cervical cancer and its precursor lesions, cervical intraepithelial neoplasia (CIN), represents a significant public health problem,induced by persistent infection of human papillomavirus (HPV). It is known that a significant percentage of CIN regresses spontaneously and only a minority of these lesions progress to cervical cancer. CIN-II is an intermediate state that can regress to CIN-I or less, or progress to CIN-III spontaneously. The rate of spontaneous regression and progression in follow-up studies are around 40-60% and 10-20%, respectively. Overestimating CIN-II lesions may cause overtreatment by excisional treatment and increase the risk of subsequent obstetric complications.

Patients newly diagnosed with CIN-II colposcopy-directed biopsy who agreed to follow up at four months intervals for at least 12 months with cervical cytology and colposcopy, were prospectively recruited. p16, ki-67 and NK receptors expression were analyzed in all CIN-II biopsies. Total regression, partial regression, persistence and progression rates of CIN-II were defined as a final outcome.

ELIGIBILITY:
Inclusion Criteria:

* preferred expectant management than immediate treatment
* exocervical histological diagnosis of CIN-II
* lesion completely visualized by colposcopy
* entire squamocolumnar junction of the cervix was visible
* showing no evidence of any immunodeficiency disease
* no history of previous cervical treatment
* could be followed-up every four months during one year
* signed consent form

Exclusion Criteria:

* not coming to follow up appointments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females with CIN-II lesion on cervical biopsy that agree to a conservative management during a period not more than 24 months, referred to the low genital tract diseases clinic of Hospital del Mar.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Status of cervix pathology using cervical smear test (CIN grade) | 2 years
  Cervical cytology test and colposcopy every 4 months starting with diagnose CIN-II or CIN-III means presence of lesion, CIN-I is regression of the lesion, and Negative is abscence of lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Mancebo, PhD, Principal Investigator — Parc de Salut Mar; Ramon Carreras, PhD, Study Chair — Parc de Salut Mar

REFERENCES:
- [Background] Discacciati MG, de Souza CA, d'Otavianno MG, Angelo-Andrade LA, Westin MC, Rabelo-Santos SH, Zeferino LC. Outcome of expectant management of cervical intraepithelial neoplasia grade 2 in women followed for 12 months. Eur J Obstet Gynecol Reprod Biol. 2011 Apr;155(2):204-8. doi: 10.1016/j.ejogrb.2010.12.002. Epub 2010 Dec 28. PMID 21193261
- [Background] Tsoumpou I, Arbyn M, Kyrgiou M, Wentzensen N, Koliopoulos G, Martin-Hirsch P, Malamou-Mitsi V, Paraskevaidis E. p16(INK4a) immunostaining in cytological and histological specimens from the uterine cervix: a systematic review and meta-analysis. Cancer Treat Rev. 2009 May;35(3):210-20. doi: 10.1016/j.ctrv.2008.10.005. Epub 2009 Mar 3. PMID 19261387
- [Background] del Pino M, Garcia S, Fuste V, Alonso I, Fuste P, Torne A, Ordi J. Value of p16(INK4a) as a marker of progression/regression in cervical intraepithelial neoplasia grade 1. Am J Obstet Gynecol. 2009 Nov;201(5):488.e1-7. doi: 10.1016/j.ajog.2009.05.046. Epub 2009 Aug 15. PMID 19683687
- [Background] Galgano MT, Castle PE, Atkins KA, Brix WK, Nassau SR, Stoler MH. Using biomarkers as objective standards in the diagnosis of cervical biopsies. Am J Surg Pathol. 2010 Aug;34(8):1077-87. doi: 10.1097/PAS.0b013e3181e8b2c4. PMID 20661011
- [Background] Guedes AC, Brenna SM, Coelho SA, Martinez EZ, Syrjanen KJ, Zeferino LC. p16(INK4a) Expression does not predict the outcome of cervical intraepithelial neoplasia grade 2. Int J Gynecol Cancer. 2007 Sep-Oct;17(5):1099-103. doi: 10.1111/j.1525-1438.2007.00899.x. Epub 2007 Mar 15. PMID 17367324
- [Background] McAllum B, Sykes PH, Sadler L, Macnab H, Simcock BJ, Mekhail AK. Is the treatment of CIN 2 always necessary in women under 25 years old? Am J Obstet Gynecol. 2011 Nov;205(5):478.e1-7. doi: 10.1016/j.ajog.2011.06.069. Epub 2011 Jun 25. PMID 21872201